CLINICAL TRIAL: NCT06563128
Title: Evaluation of the Clinical Success of Single Colour Universal Resin Composites
Brief Title: Clinical Success of Single-Color Universal Resin Composites
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mustafa Cadirci, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TDH-2023-13250
Record Dates: First submitted 2024-08-17; First posted 2024-08-20 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Dental Caries Class II

STUDY DESIGN:
Intervention Model Description: Five groups with a control goup
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Clearfil Majesty Posterior (Placebo Comparator): It is a type of composite used in the back group of teeth. It was used for the control group.
  Interventions: Other: Clearfil Majesty Posterior
- Omnichroma Universal Group (Experimental): It is a single-color universal resin composite used in both anterior and posterior group teeth.
  Interventions: Other: Omnichroma Universal Group
- Zen Universal Group (Experimental): It is a single-color universal resin composite used in both anterior and posterior group teeth.
  Interventions: Other: Zen Universal Group
- Vittra Aps Unique Universal Group (Experimental): It is a single-color universal resin composite used in both anterior and posterior group teeth.
  Interventions: Other: Vittra Aps Unique Universal Group
- Charisma Diamond Universal Group (Experimental): It is a single-color universal resin composite used in both anterior and posterior group teeth.
  Interventions: Other: Charisma Diamond Universal Group

INTERVENTIONS:
Other: Clearfil Majesty Posterior — After filling the teeth of the patients with 4 different universal resins and 1 conventional composite resin, the filling will be evaluated and recorded according to the clinical success criteria at the beginning. Then, the patients will be called back to the clinic after 6 months and 12 months, respectively, and the fillings made according to the same criteria will be re-evaluated and recorded.
  Arms: Clearfil Majesty Posterior
Other: Omnichroma Universal Group — After filling the teeth of the patients with 4 different universal resins and 1 conventional composite resin, the filling will be evaluated and recorded according to the clinical success criteria at the beginning. Then, the patients will be called back to the clinic after 6 months and 12 months, respectively, and the fillings made according to the same criteria will be re-evaluated and recorded.
  Arms: Omnichroma Universal Group
Other: Zen Universal Group — After filling the teeth of the patients with 4 different universal resins and 1 conventional composite resin, the filling will be evaluated and recorded according to the clinical success criteria at the beginning. Then, the patients will be called back to the clinic after 6 months and 12 months, respectively, and the fillings made according to the same criteria will be re-evaluated and recorded.
  Arms: Zen Universal Group
Other: Vittra Aps Unique Universal Group — After filling the teeth of the patients with 4 different universal resins and 1 conventional composite resin, the filling will be evaluated and recorded according to the clinical success criteria at the beginning. Then, the patients will be called back to the clinic after 6 months and 12 months, respectively, and the fillings made according to the same criteria will be re-evaluated and recorded.
  Arms: Vittra Aps Unique Universal Group
Other: Charisma Diamond Universal Group — After filling the teeth of the patients with 4 different universal resins and 1 conventional composite resin, the filling will be evaluated and recorded according to the clinical success criteria at the beginning. Then, the patients will be called back to the clinic after 6 months and 12 months, respectively, and the fillings made according to the same criteria will be re-evaluated and recorded.
  Arms: Charisma Diamond Universal Group

SUMMARY:
According to FDI criteria, the success of 4 different universal resin composites was targeted. In our study, a total of 180 teeth will be restored in class 2 cavities with 5 different composite resins in 5 groups.

DETAILED DESCRIPTION:
The study will be conducted in the clinic of the Atatürk University Faculty of Dentistry, Department of Restorative Dental Treatment. After the participants fulfil the inclusion criteria, no interventional procedures other than the treatments routinely applied in the clinic will be performed. Participants who apply to the clinic with the need for dental caries treatment will be included in the study if they accept it. Before the treatment, anamnesis will be taken from the participants, and their information (age, gender) will be recorded. If necessary, local anaesthesia will be applied before or after opening the cavity. If anaesthesia is applied, they will be asked whether they feel numbness. In the study, a total of 180 teeth in 5 groups will be restored with 5 different composite resins.

Group 1: Omnichroma Group 2: Vittra Aps Unique Group 3: OneShade Group 4: Charisma Diamond Group 5: Clearfil Majesty Posterior

Then, the cavity will be prepared by using diamond rond and steel rond drills in class 2 cavity preparation. After the enamel surfaces of the teeth are roughened and washed with 37% orthophosphoric acid for 30 seconds, the necessary isolation will be provided with cotton pellets and saliva absorbent. Teeth will be fixed with matrix band and wedge systems. The adhesive bond system will be applied to all surfaces of the cavity with a bonding brush according to the manufacturer's instructions. Air will be gently applied to the cavity surface to create a shiny surface with an air gun. It will then be polymerised with an LED light device. Next, five different resin composites will be placed in the respective cavities and polymerised again with the light device. Finishing operations will be performed with a diamond-lobed milling cutter, and polishing operations will be performed with rubber systems. To evaluate the clinical success of the restorations, participants will be called at 1 week (baseline), 6 months, and 1 year to be evaluated by two specialists using FDI criteria and the results will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* The patient should not have any systemic disease.
* You must be 18 years of age or older.
* The patient must have good periodontal health.
* Must have acceptable oral hygiene.
* The teeth to be restored must be symptom-free and vital.
* The mesial and distal surfaces of the teeth to be restored must be in contact with the proximal teeth.
* The tooth to be restored must be in occlusion with its antagonist.
* The tooth to be restored must have a class 2 caries lesion radiographically not exceeding 2/3 of the dentin.
* Patients with caries have an ICDAS 3-4 score.
* Voluntary acceptance to participate in the study after being informed about the study.

Exclusion Criteria:

* The patient has any systemic disease.
* Previously adhered restoration and endodontic treatment on the tooth to be restored.
* Poor periodontal health of the patient.
* Poor oral hygiene.
* The patient is pregnant or breastfeeding.
* The patient is undergoing orthodontic treatment.
* The patient has bruxism (tooth clenching) and a dry mouth.
* The teeth are devitalised.
* The patient refused to participate in the study after being informed about the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-08-27 (Actual); Study Completion 2025-11-27 (Estimated)

PRIMARY OUTCOMES:
Group 1: Omnichroma (Tokuyama Dental) Universal Composite | Baseline, 6th month and 12th month
  Restorations will be assessed at baseline, 6 months, and 12 months by two pre-calibrated and experienced dentists who are blinded to the restorative material used. The evaluations will be performed according to FDI and modified USPHS criteria. In cases of discrepancies between the assessors, the restorations will be re-evaluated by both assessors, and a final consensus will be reache.
Group 2: Vittra APS Unique (FGM) Universal Composite | Baseline, 6th month and 12th month
  Restorations will be assessed at baseline, 6 months, and 12 months by two pre-calibrated and experienced dentists who are blinded to the restorative material used. The evaluations will be performed according to FDI and modified USPHS criteria. In cases of discrepancies between the assessors, the restorations will be re-evaluated by both assessors, and a final consensus will be reache.
Group 3: Zen Chroma (President Dental) Universal Composite | Baseline, 6th month and 12th month
  Restorations will be assessed at baseline, 6 months, and 12 months by two pre-calibrated and experienced dentists who are blinded to the restorative material used. The evaluations will be performed according to FDI and modified USPHS criteria. In cases of discrepancies between the assessors, the restorations will be re-evaluated by both assessors, and a final consensus will be reache.
Group 4: Charisma Diamond (Kulzer) Universal Composite | Baseline, 6th month and 12th month
  Restorations will be assessed at baseline, 6 months, and 12 months by two pre-calibrated and experienced dentists who are blinded to the restorative material used. The evaluations will be performed according to FDI and modified USPHS criteria. In cases of discrepancies between the assessors, the restorations will be re-evaluated by both assessors, and a final consensus will be reache.
Group 5: Clearfill Majesty Posterior (Kuraray) Dental Composite | Baseline, 6th month and 12th month
  Restorations will be assessed at baseline, 6 months, and 12 months by two pre-calibrated and experienced dentists who are blinded to the restorative material used. The evaluations will be performed according to FDI and modified USPHS criteria. In cases of discrepancies between the assessors, the restorations will be re-evaluated by both assessors, and a final consensus will be reache.

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Çadırcı, Study Director — Atatürk University Faculty of Dentistry Research Assistant
Locations (1):
- Ataturk University Faculty of Dentistry Department of Restorative Dentistry Clinic, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No